CLINICAL TRIAL: NCT07141940
Title: The Role of Indonesian-Language Application-Based Auditory Guided Imagery Therapy on The Reduction of Insomnia Severity Index and Fasting Blood Glucose Levels in Diabetic Patients With Insomnia
Brief Title: Indonesian-Language Application-Based Guided Imagery Therapy for Insomnia and Glycemic Control in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Rudi Putranto, Dr. dr. Rudi Putranto, Sp.PD, K-P.P.M, MPH, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSCM_IPD_PPM_2025.01
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-03

CONDITIONS: Diabetes (Insulin-requiring, Type 1 or Type 2); Insomnia Type; Sleep Disorder; Fasting Plasma Glucose
Keywords: guided imagery; relaxation therapy; psycoeducation; insomnia; sleep disorders; fasting blood glucose; diabetes mellitus; Indonesian-language; application-based
MeSH Terms: conditions — Diabetes Mellitus; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The participants receive psychoeducation at the enrollment. Then, they were asked to use the Indonesian-language application-based auditory guided imagery therapy 3 times a week for 4 weeks.
  Interventions: Other: Indonesian-language application-based auditory guided imagery therapy
- Control Group (Active Comparator): The participants receive only psychoeducation at the enrollment.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: Indonesian-language application-based auditory guided imagery therapy — This study used a mobile application developed by researchers using Indonesian language to deliver an auditory guided imagery therapy
  Arms: Intervention Group
Other: Psychoeducation — Psychoeducation consists of sleep hygiene and relaxation therapy (breathing exercise, progressive muscle relaxation, and guided imagery)
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if guided imagery therapy using mobile application in Indonesian language can improve sleep quality and lower fasting blood glucose levels in diabetics patients who have problems with their sleep.

The main questions it aims to answer are:

* Can the app-based guided imagery therapy help improve sleep quality in diabetic patients who have trouble sleeping?
* Can the app-based guided imagery therapy help lowering fasting blood glucose in diabetic patients who have trouble sleeping? Researchers will compare app-based guided imagery therapy to education about how to sleep well, to see if the app works to improve sleep quality and lower blood glucose.

Participants will:

* Receive education about how to sleep well
* Use the app 3 times a week for 4 weeks (only for group who receive the app)
* Visit the clinic after 4 weeks for tests

ELIGIBILITY:
Inclusion Criteria:

* Patients at Endocrinology or Psychosomatic Clinic, Cipto Mangunkusumo Hospital
* Already diagnosed with Diabetes Mellitus
* HbA1c less than 12%
* Insomnia Severity Index more than 8
* Lives in Jakarta, Bogor, Depok, Tangerang, or Bekasi
* Able to understand the Indonesian language well

Exclusion Criteria:

* History of amputation or routine hemodialysis
* No device available to connect with the application
* Inability to independently access or use the application
* Inability to perform self-monitoring of blood glucose at home
* Hearing impairment
* Cognitive impairment or intellectual limitations

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | 4 weeks
Fasting Plasma Glucose | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rudi Putranto, Internist, MPH, PhD, Principal Investigator — Division of Psychosomatic and Palliative, Department of Internal Medicine, Faculty of Medicine Universitas Indonesia - Cipto Mangunkusumo Hospital
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided